CLINICAL TRIAL: NCT07243678
Title: Pharmacokinetic Assessment of Betaine Supplementation in Lactating Mothers
Acronym: BetMilkII
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PIC-142-25; PIC-142-25 (Other: Hospital Sant Joan de Déu)
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Breast Milk Fortifier Supplements
Keywords: Breast milk; Betaine; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: This is an interventional nutritional study using a within-subject design, in which lactating women receive sequential low-dose (400 milligrams/day) and high-dose (1.5 grams/day) oral betaine supplementation to assess its dynamics in breast milk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Betaine Supplementation (Sequential Low and High Dose) (Experimental): Participants will receive oral betaine supplementation at a low dose (400 milligrams/day) for one week, followed by a high dose (1.5 grams/day) for one additional week. Milk samples will be collected at baseline and at multiple time points to evaluate betaine dynamics, accumulation, and associated metabolic changes.
  Interventions: Dietary Supplement: Betaine supplement

INTERVENTIONS:
Dietary Supplement: Betaine supplement — Oral betaine supplementation will be administered to lactating women. Participants will receive a dose of 400 milligrams/day for 1 week, followed by 1.5 grams/day for an additional week.

SUMMARY:
In this study, the investigators will evaluate the dynamics of betaine excretion into breast milk following supplementation. Milk betaine concentrations will be measured at baseline (0 hours) and at 3, 6, and 12 hours after the first dose of 400 milligrams (mg) betaine to assess the short-term impact of maternal betaine supplementation on milk betaine concentration and related metabolites during 12 hours after intake. These measurements will be repeated after one week of daily supplementation with this low dose. Subsequently, the same protocol will be conducted using a higher dose (1.5 gram/day) for one additional week to compare milk betaine concentration and related metabolites before and after the supplementation period at two different doses. Depending on the outcomes, the investigators will also analyze milk macronutrient composition and explore untargeted metabolomic changes.

ELIGIBILITY:
Inclusion Criteria:

* Exclusively breastfeeding
* Infant age between 2 and 5 months

Exclusion Criteria:

* Multiple pregnancy
* Infant weight at recruitment < -1 standard deviations (SD)
* Cystathionine Beta-Synthase (CBS) deficiency (inherited disease)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Baseline, 1 week, 2 weeks
  Treatment safety and tolerability will be evaluated by assessing differences in the incidence of potential adverse events, focusing on gastrointestinal symptoms.
Change in betaine concentration in human milk | Baseline (0, 3, 6, 12 hours), 1 week (0, 3, 6, 12 hours), 2 weeks (0, 3, 6, 12 hours)
  Variation in betaine levels in breast milk measured at baseline (0 hours) and at 3 hours, 6 hours, and 12 hours after taking supplement

SECONDARY OUTCOMES:
Changes in the one-carbon metabolite profile of breast milk | Baseline (0, 3, 6, 12 hours), 1 week (0, 3, 6, 12 hours), 2 weeks (0, 3, 6, 12 hours)
  Milk samples will be analyzed by liquid chromatography-mass spectrometry to quantify betaine-related metabolites, including dimethylglycine, methionine, S-adenosylmethionine, S-adenosylhomocysteine, cystathionine, choline, homocysteine, methyl folate, and folic acid at the different time-points.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sant Joan de Deu, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No